CLINICAL TRIAL: NCT00321633
Title: A Randomized Phase II Pilot Trial of Carboplatin Compared to Docetaxel for Patients With Metastatic Genetic Breast Cancer [BRCA Trial]
Brief Title: Carboplatin or Docetaxel in Treating Women With Metastatic Genetic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University College London Hospitals (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000467994; CRUK-BRCA-TRIAL; EUDRACT-2004-001496-20; EU-20603; ISRCTN43372330; BBC-CRUK-BRCA-TRIAL
Record Dates: First submitted 2006-05-02; First posted 2006-05-04 (Estimated); Last update posted 2013-08-26 (Estimated); Status verified 2009-07

CONDITIONS: brca1 Mutation Carrier; brca2 Mutation Carrier; Breast Cancer; Hereditary Breast/Ovarian Cancer (brca1, brca2)
Keywords: stage IV breast cancer; recurrent breast cancer; hereditary breast/ovarian cancer (BRCA1, BRCA2); BRCA1 mutation carrier; BRCA2 mutation carrier
MeSH Terms: conditions — Breast Neoplasms; Hereditary Breast and Ovarian Cancer Syndrome | interventions — Carboplatin; Docetaxel

INTERVENTIONS:
Drug: carboplatin
Drug: docetaxel

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as carboplatin and docetaxel, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. It is not yet known whether carboplatin is more effective than docetaxel in treating patients with metastatic genetic breast cancer.

PURPOSE: This randomized phase II trial is studying carboplatin to see how well it works compared to docetaxel in treating women with metastatic genetic breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the safety and effectiveness of carboplatin vs docetaxel in women with metastatic breast cancer and the BRCA1 or BRCA2 gene mutation.

Secondary

* Compare time to disease progression in patients treated with these regimens.
* Compare progression-free survival of patients treated with carboplatin vs docetaxel.

OUTLINE: This is a randomized, open-label, multicenter, pilot study. Patients are stratified according to gene mutation (BRCA1 vs BRCA2), prior adjuvant taxane chemotherapy (yes vs no), liver or lung metastasis affecting the parenchyma (yes vs no), Jewish ancestry by parent or grandparent (yes vs no), and first-line treatment vs second-line treatment. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive carboplatin IV over 1 hour on day 1.
* Arm 2: Patients receive docetaxel IV over 1 hour on day 1. In both arms, treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity. Patients with disease progression after 3 or 6 courses of treatment may crossover to the alternative treatment arm. If progression is present after 3 courses in the crossover arm, patients may receive further treatment at the discretion of their oncologist. Patients responding to and tolerating treatment well, may be given 2 further courses in accordance with local center policy, although this is not encouraged.

Patients with HER2-positive disease may receive trastuzumab (Herceptin®) IV once every 7 or 21 days.

After completion of study treatment, patients are followed periodically for survival.

Peer Reviewed and Funded or Endorsed by Cancer Research UK

PROJECTED ACCRUAL: A total of 148 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed breast cancer

  * BRCA1 or BRCA2 mutation carrier
  * Metastatic disease
* Measurable disease, defined as ≥ 1 unidimensionally measurable lesion ≥ 20 mm by conventional techniques or ≥ 10 mm by spiral CT scan
* Stable, treated brain metastases allowed provided other sites of measurable disease are present
* Patients with bone metastases who are currently receiving bisphosphonates for palliation are eligible provided other sites of measurable disease are present
* Patients who have not received anthracycline-based chemotherapy in the adjuvant setting may receive a non-taxane, anthracycline regimen as the first-line metastatic treatment and enter the trial at confirmed progression (second-line)
* No bone-limited disease
* No disease suitable for endocrine therapy alone
* Hormone receptor status not specified

PATIENT CHARACTERISTICS:

* Menopausal status not specified
* Sex: female
* WHO performance status 0-2
* Life expectancy ≥ 3 months
* AST and/or ALT ≤ 5 times upper limit of normal (ULN) (≤ 3 if alkaline phosphatase > 5 times ULN)
* Glomerular filtration rate ≥ 30 mL/min
* Normal urea and creatinine
* Normal hematological and biochemical studies
* Normal bilirubin
* Not pregnant or nursing
* Fertile patients must use effective contraception during and for 6 months after completion of study treatment
* Negative pregnancy test
* No known allergy to platinum compounds or mannitol
* No known sensitivity to taxanes
* No other malignancy within the past 10 years except adequately treated in situ carcinoma of the cervix or basal cell or squamous cell carcinoma of the skin
* No sensory or motor neuropathy > grade 1
* No other serious uncontrolled medical conditions or concurrent medical illness that would preclude study compliance
* No contraindication to chemotherapy

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* At least 12 months since prior taxane therapy
* No prior chemotherapy with a platinum drug, unless treatment was for a non-breast cancer-related disease more than 10 years ago

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 148 (Estimated)
Dates: Start 2005-09; Primary Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Response and toxicity

SECONDARY OUTCOMES:
Time to progression

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Tutt, MD, PhD, FRCR, MBBS, MRCP, Study Chair — Guy's Hospital
Locations (25):
- Royal Melbourne Hospital, Parkville, Victoria, Australia
- Israel (3):
  - Soroka University Medical Center, Beersheba
  - Naharia Hospital, Nahariya
  - Chaim Sheba Medical Center, Tel Litwinsky
- Instituto Portugues de Oncologia de Francisco Gentil - Centro Regional de Oncologia de Lisboa, SA, Lisbon, Portugal
- Vall d'Hebron University Hospital, Barcelona, Spain
- Lund University Hospital, Lund, Sweden
- United Kingdom (18):
  - Addenbrooke's Hospital, Cambridge, England
  - Royal Devon and Exeter Hospital, Exeter, England
  - UCL Cancer Institute, Hampstead, London, England
  - Cookridge Hospital, Leeds, England
  - Leeds Cancer Centre at St. James's University Hospital, Leeds, England
  - Guy's Hospital, London, England
  - Royal Marsden - Surrey, London, England
  - Christie Hospital, Manchester, England
  - Clatterbridge Centre for Oncology, Merseyside, England
  - James Paget Hospital, Norfolk, England
  - Mount Vernon Cancer Centre at Mount Vernon Hospital, Northwood, England
  - Norfolk and Norwich University Hospital, Norwich, England
  - Dorset Cancer Centre, Poole Dorset, England
  - Portsmouth Oncology Centre at Saint Mary's Hospital, Portsmouth Hants, England
  - Southampton General Hospital, Southampton, England
  - Torbay Hospital, Torquay, England
  - Edinburgh Cancer Centre at Western General Hospital, Edinburgh, Scotland
  - Velindre Cancer Center at Velindre Hospital, Cardiff, Wales